CLINICAL TRIAL: NCT00049946
Title: A Multicenter, Double-Blind, Double-Dummy, Placebo-Controlled, Randomized, Parallel Group Evaluation of the Efficacy and Safety of a Fixed-Dose of Talnetant Versus Placebo Versus Risperidone in Subjects With Schizophrenia
Brief Title: Schizophrenia Study In Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SB223412/078
Record Dates: First submitted 2002-11-15; First posted 2002-11-18 (Estimated); Last update posted 2017-08-16 (Actual); Status verified 2017-08

CONDITIONS: Schizophrenia
Keywords: Talnetant; schizophrenia; NK3 receptor antagonist; psychosis
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — SB 223412; Risperidone

INTERVENTIONS:
Drug: talnetant
Drug: risperidone

SUMMARY:
A Placebo Controlled Study For Patients With Schizophrenia

ELIGIBILITY:
Inclusion Criteria:

* Patient must meet diagnostic criteria for schizophrenia.

Exclusion Criteria:

* Patients with other psychotic disorders.
* Patients whose condition is due to the direct physiological effects of a substances (e.g., drug abuse) or a general medical condition.
* Patients with a history of autistic disorder or another pervasive developmental disorder.
* Patients with epilepsy or a history of seizures requiring treatment.
* Patients who are excluded from taking the drug risperidone.
* Patients who pose a current serious suicidal or homicidal risk.
* Patients who are adequately stabilized on their treatment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 231
Dates: Start 2002-10; Primary Completion 2003-04 (Actual); Study Completion 2003-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the PANSS total score.

SECONDARY OUTCOMES:
Secondary measures assessed efficacy, safety & tolerability endpoints using the PANSS, BPRS Psychosis score, CGI-S, CGI-GI, Calgary Depression Scale for Schizophrenia, Brief Assessment of Cognition for Schizophrenia, and others.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, MD, Study Director — GlaxoSmithKline
Locations (30):
- United States (30):
  - GSK Clinical Trial Call Center, Scottsdale, Arizona
  - GSK Clinical Trial Call Center, Cerritos, California
  - GSK Clinical Trial Call Center, Chula Vista, California
  - GSK Clinical Trial Call Center, Garden Grove, California
  - GSK Clinical Trial Call Center, Orange, California
  - GSK Clinical Trial Call Center, Pico Rivera, California
  - GSK Clinical Trial Call Center, Rosemead, California
  - GSK Clinical Trial Call Center, Sacramento, California
  - GSK Clinical Trial Call Center, San Diego, California
  - GSK Clinical Trial Call Center, New Britain, Connecticut
  - GSK Clinical Trial Call Center, New Haven, Connecticut
  - GSK Clinical Trial Call Center, Washington D.C., District of Columbia
  - GSK Clinical Trial Call Center, North Miami, Florida
  - GSK Clinical Trial Call Center, Tampa, Florida
  - GSK Clinical Trial Call Center, Winter Park, Florida
  - GSK Clinical Trial Call Center, Hoffman Estates, Illinois
  - GSK Clinical Trial Call Center, Greenwood, Indiana
  - GSK Clinical Trial Call Center, Shreveport, Louisiana
  - GSK Clinical Trial Call Center, Clementon, New Jersey
  - GSK Clinical Trial Call Center, Hollis, New York
  - GSK Clinical Trial Call Center, Butner, North Carolina
  - GSK Clinical Trial Call Center, Raleigh, North Carolina
  - GSK Clinical Trial Call Center, Cincinnati, Ohio
  - GSK Clinical Trial Call Center, Cleveland, Ohio
  - GSK Clinical Trial Call Center, Norman, Oklahoma
  - GSK Clinical Trial Call Center, Oklahoma City, Oklahoma
  - GSK Clinical Trial Call Center, Nashville, Tennessee
  - GSK Clinical Trial Call Center, Austin, Texas
  - GSK Clinical Trial Call Center, Bellaire, Texas
  - GSK Clinical Trial Call Center, Terrell, Texas